CLINICAL TRIAL: NCT01065571
Title: Effects of Carrageenan-Elimination Diet on Ulcerative Colitis Disease Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: The Broad Foundation (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Joanne Kramer Tobacman, Associate Professor of Clinical Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2009-0073
Record Dates: First submitted 2010-02-04; First posted 2010-02-09 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Ulcerative Colitis
Keywords: relapse; carrageenan; inflammation
MeSH Terms: conditions — Colitis, Ulcerative; Recurrence; Inflammation | interventions — Carrageenan; Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carrageenan-free diet with placebo (Experimental): This is the experimental arm in which subjects will be on a no-carrageenan diet and receive placebo capsules. This will test whether the no carrageenan diet leads to longer relapse-free interval for patients with ulcerative colitis.
  Interventions: Other: dietary intervention with no-carrageenan diet
- carrageenan-free diet w/ carrageenan (Active Comparator): The carrageenan-free diet with carrageenan supplement will mimic the carrageenan normally consumed in the diet. The study will permit blinded comparison of carrageenan-free vs. carrageenan consumption.
  Interventions: Dietary Supplement: carrageenan

INTERVENTIONS:
Dietary Supplement: carrageenan — The intervention is the carrageenan-free diet. Supplementary carrageenan capsules will be given to mimic the carrageenan in the normal diet.
  Arms: carrageenan-free diet w/ carrageenan
Other: dietary intervention with no-carrageenan diet — The intervention will consist of the no-carrageenan diet.
  Arms: carrageenan-free diet with placebo

SUMMARY:
The study hypothesis is that withdrawal of carrageenan will lead to a longer, relapse free interval in patients with ulcerative colitis.

DETAILED DESCRIPTION:
This study will evaluate the interval to relapse in patients with ulcerative colitis. The patients will be adults, who have been in remission for at least one month. They will have previously required corticosteroids to induce remission. Subjects will be instructed in a no-carrageenan diet and required to follow this diet for the duration of their participation in the clinical study. They will be randomized to receive either placebo capsules or capsules containing carrageenan 100 mg. In this way, the study will be a double blind study of no-carrageenan vs. carrageenan. Main study outcome is the interval to relapse. Since ulcerative colitis is associated with relapses, relapse is anticipated. Other outcome measures will include scores on questionnaires, including the SSCAI and the SIDBQ, and laboratory measurements of inflammation.

Subjects will participate for one year or until relapse, with study visits every three months and telephone contacts every two weeks. After three months, participants will increase to two capsules daily, of either placebo or carrageenan.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis
* Adult
* In remission
* Required corticosteroids to induce remission
* Able to make food choices and follow diet

Exclusion Criteria:

* Not able to make food choices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Tobacman, M.D., Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carrageenan-free Diet With Placebo | Carrageenan-free Diet w/ Carrageenan
Started | 10 | 5
Completed | 7 | 5
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carrageenan-free Diet With Placebo | Carrageenan-free Diet w/ Carrageenan | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (5) | 54 (5) | 51 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Relapses by Group
Description: log-rank test to test for difference in number of relapses by group
Time Frame: up to one year of participation for each enrolled subject
Measure: Number; unit: relapses
Arm/Group | Carrageenan-free Diet With Placebo | Carrageenan-free Diet w/ Carrageenan
Number analyzed (Participants) | 7 | 5
relapses | 0 | 3
Statistical Analysis 1: Comparison: Carrageenan-free Diet With Placebo vs Carrageenan-free Diet w/ Carrageenan; Kaplan-Meier life table analysis was performed to compare the two groups. The null hypothesis was that there would be no difference in relapses between the two groups during the study; Test type: Equivalence — Non-parametric analysis of interval to relapse; p = 0.046, Log Rank — result from log rank test

2. Secondary Outcome: Fecal Calprotectin (Microgram/Gram Stool)
Description: paired t-test comparing mean values at baseline and at end of study participation by group
Time Frame: one year or relapse or withdrawal compared with baseline
Population: participants who had fecal calprotectin tests at baseline and at end of participation at one year or at time of relapse or withdrawal from study participation
Measure: Mean (Standard Deviation); unit: micrograms/gm stool
Arm/Group | Carrageenan-free Diet With Placebo | Carrageenan-free Diet w/ Carrageenan
Number analyzed (Participants) | 5 | 5
micrograms/gm stool | -18.4 (170) | 37.8 (33)
Statistical Analysis 1: Comparison: Carrageenan-free Diet With Placebo vs Carrageenan-free Diet w/ Carrageenan; Test type: Superiority — fecal calprotectin (micrograms/gm stool); p = 0.06, t-test, 2 sided

3. Secondary Outcome: Serum Interleukin-6 (pg/ml)
Description: Difference in IL-6 between groups between baseline and end of study participation
Time Frame: change in IL-6 between baseline and up to one year of study participation
Population: change in IL-6 between baseline and end of participation
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- no Carrageenan Group: carrageenan-free diet with placebo group
- Carrageenan Exposed: carrageenan-free diet with added carrageenan group
Arm/Group | no Carrageenan Group | Carrageenan Exposed
Number analyzed (Participants) | 4 | 5
pg/ml | -1.11 (2.22) | 2.44 (1.49)
Statistical Analysis 1: Comparison: no Carrageenan Group vs Carrageenan Exposed; paired t-test comparing baseline and value at end of participation; Test type: Superiority; p = 0.02, t-test, 2 sided — not adjusted for muliple comparisons, a priori threshold of 0.05

ADVERSE EVENTS:
Arm/Group | Carrageenan-free Diet w/ Carrageenan | Carrageenan-free Diet With Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No